CLINICAL TRIAL: NCT02317081
Title: Axetis Inert Coronary Stent System First In Man Clinical Investigation (AXETIS FIM)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Axetis AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AXETIS FIM
Record Dates: First submitted 2014-11-19; First posted 2014-12-15 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Native Coronary Artery Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axetis Inert Coronary Stents (Experimental): Axetis Inert Coronary Stents for de novo coronary lesion
  Interventions: Device: Axetis Inert Coronary Stents

INTERVENTIONS:
Device: Axetis Inert Coronary Stents — de novo coronary artery stenosis in native vessels

SUMMARY:
Prospective, multicenter, single arm study, to assess the feasibility and safety of the Axetis Inert Stent for treatment of patients with de novo coronary artery stenosis in native vessels.

DETAILED DESCRIPTION:
Prospective, multicenter, open-label and single arm study, conducted in 3 interventional cardiology centers in The Netherlands. The objective is to assess the feasibility and safety of the Axetis Inert Stent for treatment of patients with de novo coronary artery stenosis in native vessels. In total, 35 patients will be enrolled. All patients will be treated with Axetis Inert Coronary Stent System. All patients will undergo repeat angiography at 6 months follow-up. Quantitative coronary angiography (QCA) assessment will be performed at baseline (pre- and post-procedure) and at 6 months follow-up. All patients will undergo Optical coherence Tomography (OCT) investigation at baseline (post procedure) and at 6 months follow-up. The primary endpoint is in-stent Late Lumen Loss (LLL) at 6 months after stent implantation as assessed by off-line QCA. Clinical follow-up will occur at 6 and 12 months post-stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years
* Evidence of myocardial ischemia without elevatedTroponin / cardiac biomarkers (e.g.

stable or unstable angina, silent ischemia demonstrated by positive territorial functional study). NSTEMI patients are allowed, as long as Troponin is within the normal limits before the start of the procedure.

* The patient has a planned intervention of up to two de-novo lesions in two different vessels (previously untreated vessels)
* Lesion must have a visually estimated diameter stenosis of ≥50% and <100%.
* Lesion length must be ≤ 28 mm
* RVD must be between 2.4 and 3.8 mm
* Written informed consent
* The patient and the patient's physician agree to the follow-up visits including angiographic follow-up and OCT control at 6 months

Exclusion Criteria:

* Evidence of ongoing acute myocardial infarction in ECG and or elevated cardiac biomarkers prior to procedure.
* LVEF <30%
* Platelet count <100,000 cells/mm3 or >400,000 cells/mm3, a WBC of <3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis)
* Known renal insufficiency (e.g., eGFR <60 ml/kg/m2 or serum creatinine level of >2.5 mg/dL, or subject on dialysis)
* History of bleeding diathesis or coagulopathy
* The patient is a recipient of a heart transplant
* Known hypersensitivity or contraindication to aspirin, heparin, antiplatelet medication specified for use in the study (clopidogrel, prasugrel, ticagrelor and ticlopidine) or stainless steel
* Other medical illness (e.g. cancer, stroke with neurological deficiency) or known history of substance abuse (alcohol, cocaine, heroin etc.) as per physician judgment that may cause non-compliance with the protocol or confound the data interpretation or is associated with a limited life expectancy
* Pregnant or breastfeeding woman or woman in fertile period not taking adequate contraceptives
* Severe tortuous, calcified or angulated coronary anatomy of the study vessel that in the opinion of the investigator would result in suboptimal imaging or excessive risk of complication from placement of an OCT catheter
* Target lesion in left main stem.
* Target lesion involves a side branch > 2.0mm in diameter
* Aorto-ostial target lesion (within 3 mm of the aorta junction).
* Total occlusion or TIMI flow 1, prior to wire crossing
* The target vessel contains visible thrombus
* Restenotic lesion
* Target vessel with previously placed stent or with graft
* Located within an arterial or saphenous vein graft
* Treatment of more than 1 lesion in one vessel, or treatment of more than two lesions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
In-stent Late Lumen Loss (LLL) assessed by off-line QCA | 6 months after stent implantation

SECONDARY OUTCOMES:
Acute Lumen gain | Post intervention (1 hour)
  Angiographic endpoint MLD (mm); Diameter Stenosis (%); Binary Restenosis (DS ≥50%)
Acute area gain | Post intervention (1 hour)
  Optical coherence tomography end point
Percent Acute device success | 1 day post intervention
  Device-oriented Composite Endpoints (DoCE) at 6 months and 12 months (DoCE is defined as Cardiac Death, MI not clearly attributable to a nonintervention vessel, and clinically-indicated Target Lesion Revascularization and its individual components) Stent thrombosis according to the ARC definitions up to 12 months follow-up
late lumen loss | 6 months after intervention
  Angiographic endpoint
maximal neointimal thickness | 6 months after intervention
  OCT
Percent procedural success | post intervention (1 hour)
Number of adverse cardiac events | 12 months after intervention
  clinical endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Teunissen, PhD, Study Director — Cardialysis BV; Mariann Gyöngyösi, Prof. MD, Principal Investigator — University Hospital, Cardiology, Vienna, Austria
Locations (3):
- Netherlands (3):
  - AMC Amsterdam, Netherlands, Amsterdam
  - Thoraxcentrum Twente, Medisch Spectrum, Enschede
  - St. Antonius, Nieuwegein